CLINICAL TRIAL: NCT03422055
Title: Study of Tolerance, Biodistribution and Dosimetry of Fucoidan Radiolabeled by Technetium-99m
Acronym: NANO-ATHERO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P130201J
Record Dates: First submitted 2018-01-15; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteer
Keywords: safety 99mTc-Fucoïdane scintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-Fucoidan SPECT (Experimental)
  Interventions: Drug: 99mTc-Fucoidan SPECT

INTERVENTIONS:
Drug: 99mTc-Fucoidan SPECT — Intravenous administration of 99mTc-Fucoidan on healthy volunteers.

SUMMARY:
The development of an innovative imaging agent capable of non-invasively detecting vulnerable plaques is a major objective of research in cardiovascular pathology. Such a tool would allow for better identification of patients at risk of acute events. We showed that 99mTechnetium (99mTc)-labeled fucoidan was able to target P-selectine expressed by activated platelets in vitro in humans and in vivo in a model of abdominal aortic aorta thrombus and endocarditic vegetations in rats.

One of the objectives of the Nanoathero program is the clinical translation of the 99mTc-fucoidan. As a first step, we will assess the safety, biodistribution and dosimetry of this new radiopharmaceutical in humans.

DETAILED DESCRIPTION:
The development of an innovative imaging agent capable of non-invasively detecting vulnerable plaques is a major objective of research in cardiovascular pathology. Such a tool would allow for better identification of patients at risk of acute events. We showed that 99mTechnetium-labelled fucoidan was able to target P-selectin expressed by activated platelets in vitro in humans and in vivo in a model of abdominal aortic aorta thrombus and endocarditic vegetations in rats.

NanoAthero is a monocenter, interventional, open-labeled, first-in-man study to evaluate tolerance of 99mTc-Fucoïdane in healthy volunteers.

Healthy volunteers registered in the Bichat Centre for Clinical Investigations (CCI) will be contacted by email to participate in the study. The selection visit will be organized by the CCI according to the availability of the healthy volunteer.

V0: selection/inclusion visit: pre-audit of eligibility criteria, demographic data, medical examination, clinical examination and measurement of vital signs, urinary pregnancy test for women of childbearing potential, blood samples (hematology and biochemistry analyses) and 12-lead ECG.

V1: 99mTc-Fucoidan scintigraphy. The delay between the inclusion visit and the completion of the scan is 30 ± 7 days. The visit will include verification and confirmation of the consent of the healthy volunteer, clinical examination and measurement of vital signs, urinary pregnancy test for women of childbearing age, blood samples (hematology and biochemistry analyses) and 12-lead ECG.

Whole-body scintigraphic acquisitions will be performed 30 min, 90 min, 3 hours, 6 hours and 24 hours after intravenous administration of 99mTc-Fucoidan for the evaluation of biodistribution and dosimetry. Vital signs will be monitored 5 min, 15 min, 30 min, 60 min, 90 min, 3 hours, 6 hours and 24 hours after intravenous administration of 99mTc-Fucoidan. 24-hour urine collection will be performed for dosimetry assessment.

V2: End of research visit will be carried out 7 ± 3 days after administration of 99mTc-Fucoidan, and will include medical interview, clinical examination, measurement of vital signs, blood samples (hematology and biochemistry analyses) and 12-lead ECG.

ELIGIBILITY:
Inclusion criteria :

* Adult volunteer
* No chronic progressive disease
* Absence of long term medication
* BMI between 18 and 35
* Absence of chronic infection by HIV, HVB, HCV
* Absence of significant biological abnormality in the screening report
* Affiliation to a social security system or CMU
* Signed informed consent
* Females with childbearing potential as well as males should use effective contraceptive methods

Exclusion criteria :

* Pregnant or nursing woman
* Person of exclusion period of research protocol
* Person in detention by judicial or administrative decision
* Protected person (maintenance of justice, tutelage, legal guardianship)
* Person unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events and serious adverse events after 99m Tc-Fucoidan IV administration | up to 7 days
  Number and percentage of subjects with adverse events and serious adverse events based on clinical, ECG and biological monitoring until 7 days after 99mTc-Fucoidan intravenous administration

SECONDARY OUTCOMES:
Biodistribution of 99mTc-Fucoidan after intravenous administration | during 24h after injection
Dosimetry of 99mTc-Fucoidan after intravenous administration | during 24h after injection

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Le Guludec, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Bichat - Claude Bernard, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oostveen RF, Zheng KH, Kaiser Y, Nurmohamed NS, Kroon J, de Wit TC, Poel E, Aerts J, Rouzet F, Stroes ESG, Letourneur D, Verberne HJ, Chauvierre C, Stahle MR. First-in-human study of 99mTc-labeled fucoidan, a SPECT tracer targeting P-selectin. EJNMMI Res. 2024 Nov 19;14(1):112. doi: 10.1186/s13550-024-01173-8. PMID 39562382